CLINICAL TRIAL: NCT02013869
Title: Low Flow Anaesthesia; Cost-effectiveness of the Flow-I Anaesthesia Machine, a Comparison to Established Anaesthesia Delivery Unit
Brief Title: Low Flow Anaesthesia, is There a Difference Between 2 Modern Anaesthetic Machines Using Different Gas Reservoir
Acronym: LF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Two of the sites withdraw, did not have capacity to recruit patients
Sponsor: Jan Jakobsson (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Sponsor-Investigator, Jan Jakobsson, Adj Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 201301; JJ201301 (Other Grant/Funding Number: M201301)
Record Dates: First submitted 2013-11-29; First posted 2013-12-17 (Estimated); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: General Anaesthesia
Keywords: fresh gas flow; quality of anaesthesia; minimal alveolar concentration

STUDY DESIGN:
Intervention Model Description: We studied the time to reach a MAC value for two fifferent anaesthetic machines, Flow-i versus Aisys looking at the time to reach 1 MAC desflurane
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flow-I (Experimental): Wash in of desflurane (SupraneR) in an anaesthesia machine without below, a new technique that do not have abag/reservoir that is compressed but pushes the gas into the patient. This technique uses far less of fresh gas volume. Thus lower anaesthetic gas will be consumed per hour.
  The primary outcome is the amount of anaesthetic consumed, the decrease in liquid desflurane (SupraneR) in the vaporiser of the ananesthetic machine. The vaporizer will be weighed before and after the anaesthetic to define the amount used.
  Interventions: Device: Flow-I, a modern anaesthetic machine without a bag/below/gas reservoir for compression of insufflation gas
- Asys (Active Comparator): Wash in of desflurane (Suprane) in conventional anaesthesia machine Asys, with the anaesthesia machine Asys that has a bag/reservoir that is compressed for insufflation of gas into the patient, thus it is expected that more gas will be consumed per hour.
  The primary outcome is the amount of anaesthetic consumed, the decrease in liquid desflurane (SupraneR) in the vaporiser of the ananesthetic machine. The vaporizer will be weighed before and after the anaesthetic to define the amount used.
  Interventions: Device: Asys, a anaesthetic machine with a bag/bellow for compression of gas to be insufflated

INTERVENTIONS:
Device: Flow-I, a modern anaesthetic machine without a bag/below/gas reservoir for compression of insufflation gas — Desflurane Dialed setting 18 % on the machine gas vaporized
  Arms: Flow-I
Device: Asys, a anaesthetic machine with a bag/bellow for compression of gas to be insufflated — Desflurane dialed 18% on the machine gas vaporized
  Arms: Asys

SUMMARY:
To study the Flow-I breathing circle during low flow general anaesthesia, whether this non-below system has advantages reduced time to reach Et 1MAC (minimal alveolar concentration) and lower consumption of inhaled agent

DETAILED DESCRIPTION:
Assessing whether there are clinical differences in anaesthetic performance between standard anaesthesia workstation including a below and the new Flow-I device without a below

ELIGIBILITY:
Inclusion Criteria:

ASA 1-2 patient 18 - 65 years scheduled for elective surgery

Exclusion Criteria:

ASA > 2 heart failure COPD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Time to reach 1.5 MAC (minimal alveolar concentration) Et | 1 hour
  The time needed, seconds, to increase the end tidal desflurane concentration during wash-in from a 1 MAC to a 1.5 MAC with a constant fresh gas flow of 1 L/min and the vaporiser set a 3 MAC ( minimal alveolar concentration) (18%) will be compared between the two study groups

SECONDARY OUTCOMES:
amount of inhaled agent consumed ml/min | 5 hours
  The vaporiser will be weighed before and after each case and the amount of vapor, desflurane, consumed during the anaesthesia will be calculated Gr/min.
Postoperative Quality of Recovery | 72 hours
  Quality of recovery will be followed during the first 72 hours after anaesthesia

OTHER OUTCOMES:
Adequate anaesthesia | 5 hours
  Patients will be asked after end of anaesthesia if they have had any recall of intraoperative events

CONTACTS AND LOCATIONS:
Overall Officials: Jan g Jakobsson, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Danderyds Hospital, Stockholm, Sweden

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-11-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT02013869/Prot_SAP_000.pdf